CLINICAL TRIAL: NCT01191593
Title: The Efficacy of Adductor-Canal-Blockade on Pain and Morphine Consumption After Revision Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Pia Jaeger, M.D., Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM1-PJ-10; 2010-021161-71 (EudraCT Number)
Record Dates: First submitted 2010-08-30; First posted 2010-08-31 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Postoperative Pain; Knee Arthroplasty
Keywords: Adductor-Canal-Blockade; postoperative pain; US-guided nerve block; revision knee arthroplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adductor-Canal-Blockade with ropivacaine (Experimental)
  Interventions: Procedure: Adductor-Canal-Blockade with Ropivacaine
- Adductor-Canal-blockade with saline (Placebo Comparator)
  Interventions: Procedure: Adductor-Canal-blockade with saline

INTERVENTIONS:
Procedure: Adductor-Canal-Blockade with Ropivacaine — US-guided Adductor-Canal-Blockade with ropivacaine 7,5 mg/ml
  Other Names: Naropine; Postoperative pain; US-guided nerve block
  Arms: Adductor-Canal-Blockade with ropivacaine
Procedure: Adductor-Canal-blockade with saline — US-guided Adductor-Canal-blockade with saline
  Other Names: Placebo block
  Arms: Adductor-Canal-blockade with saline

SUMMARY:
The purpose of this study is to determine whether Adductor-Canal-Blockade is effective at reducing pain and morphine consumption after revision knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Revision Knee Arthroplasty in general anaesthesia
* American society of anesthesiologists (ASA) 1-3
* BMI 18-40
* Written informed consent

Exclusion Criteria:

* Can not cooperate to the exam
* Do not speak or understand Danish
* Drug allergy
* Alcohol or drug abuse

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Pain during 45 degrees active flexion of the knee | 4 hours postoperative
  0-100 mm at a visual analogue scale (VAS), at 4 hours postoperative.

SECONDARY OUTCOMES:
Pain during 45 degrees active flexion of the knee | 1-8 hours postoperative
  0-100 mm at a visual analogue scale (VAS), registered at the intervals 1, 2, 4, 6 and 8 hours postoperative, calculated as "the area under the curve" (AUC) for the interval 1-8 hours postoperative.
Pain during 45 degrees active flexion of the knee | 24 hours postoperative
  0-100 mm at a visual analogue scale (VAS), at 24 hours postoperative.
Pain during rest | 1-8 hours postoperative
  0-100 mm at a visual analogue scale (VAS), registered at the intervals 1, 2, 4, 6 and 8 hours postoperative, calculated as "the area under the curve" (AUC) for the interval 1-8 hours postoperative.
Pain during rest | 24 hours postoperative
  0-100 mm at a visual analogue scale (VAS), at 24 hours postoperative.
Total morphine consumption | 0-24 hours postoperative
  Total morphine consumption at the intervals 0-8, 8-24 and 0-24 hours postoperative.
Postoperative nausea | 1-8 hours postoperative
  Nausea scores(0-3)registered at 1,2,4,6 and 8 hours postoperative, calculated as mean value for the interval 1-8 hours postoperative.
Postoperative nausea | 24 hours postoperative
  Nausea score(0-3)at 24 hours postoperative.
Postoperative vomiting | 0-24 hours postoperative
  Number of vomiting episodes at the intervals 0-8, 8-24 and 0-24 hours postoperative.
Zofran consumption | 0-24 hours postoperative
  Total zofran consumption at the intervals 0-8, 8-24 and 0-24 hours postoperative.
Sedation | 1-8 hours postoperative
  Sedation score (0-3) registered at 1,2,4,6 and 8 hours postoperative, calculated as the mean value for the interval 1-8 hours postoperative.
Sedation | 24 hours postoperative
  Sedation score (0-3) at 24 hours postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Pia Jæger, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Anaesthesia and Surgery, HOC, Rigshospitalet, Denmark, Copenhagen, København Ø, Denmark

REFERENCES:
- [Derived] Jaeger P, Koscielniak-Nielsen ZJ, Schroder HM, Mathiesen O, Henningsen MH, Lund J, Jenstrup MT, Dahl JB. Adductor canal block for postoperative pain treatment after revision knee arthroplasty: a blinded, randomized, placebo-controlled study. PLoS One. 2014 Nov 11;9(11):e111951. doi: 10.1371/journal.pone.0111951. eCollection 2014. PMID 25386752